CLINICAL TRIAL: NCT03197467
Title: Neoadjuvant Anti PD-1 Immunotherapy in Resectable Non-small Cell Lung Cancer [NEOMUN]
Brief Title: Neoadjuvant Anti PD-1 Immunotherapy in Resectable Non-small Cell Lung Cancer
Acronym: NEOMUN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0316-ASG; 2016-002170-13 (EudraCT Number); MISP 52887 (Registry Identifier: MSD SHARP & DOHME GMBH)
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab at fixed dose: 200 mg q3w i.v. for 2 cycles
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab at fixed dose: 200 mg q3w i.v. for 2 cycles

SUMMARY:
NEOMUN is designed as an open-label, single arm, prospective, monocenter, phase II study of pembrolizumab in a neoadjuvant setting in patients with non-small cell lung cancer of Stage II/IIIA suitable for curative intent surgery.

DETAILED DESCRIPTION:
The study is designed as an open-label, single arm, prospective, monocenter, phase II study of pembrolizumab in a neoadjuvant setting in patients with resectable NSCLC stage II/IIIA suitable for curative intent surgery, taking place in Germany. Planned sample size is N=30.

Investigational drug is Pembrolizumab at fixed dose, given 200 mg q3w i.v. for 2 cycles. After completion of immunotherapy lobectomy/ bilobectomy with curative intent is scheduled.

Primary objectives are to assess feasibility and safety of a neoadjuvant application of pembrolizumab and to assess antitumor activity of pembrolizumab with regard to clinical and pathologic tumor response. Secondary objective is to assess the impact of neoadjuvant pembrolizumab on patient disease free and overall survival. Exploratory objective is o explore potential predictive biomarkers for pembrolizumab efficacy (immune cell imaging).

ELIGIBILITY:
Inclusion Criteria:

1. Cooperation and willingness to complete all aspects of the study
2. Signed and dated written informed consent must be given prior to study inclusion
3. Histological or cytological confirmed NSCLC
4. Clinical stage II-IIIA according to the TNM classification, 7th edition:

   stage IIIa: T1/T2 N2 (IIIa1-3 Robinson classification)
5. Adequate disease staging by PET/CT and brain MRI
6. At least 1 measurable lesion according to RECIST 1.1
7. Age ≥ 18 years
8. ECOG performance status 0 - 1
9. Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Male subjects of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
11. Adequate bone marrow function, liver and renal function:

    1. Absolute neutrophil count ≥ 1.5 x 109/L
    2. Thrombocytes ≥ 100 x 109/L
    3. Hemoglobin ≥ 9 g/dL without transfusion or EPO dependency (within 7 days of assessment)
    4. INR < 1.4 ULN and PTT < 40 seconds during the last 7 days before therapy
    5. Bilirubin < 1.5 x upper limit of normal
    6. AST (GOT) and ALT (GPT) < 2.5 x ULN
    7. Albumin >2.5 mg/dL
    8. Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl): ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
12. Adequate lung and cardiac function for intended lung resection according to German S3 guideline

Exclusion Criteria:

1. Anticancer treatment during the last 30 days prior to start of treatment, including systemic therapy, radiotherapy or major surgery
2. Participation in a clinical trial within the last 30 days prior to study treatment
3. History of allogeneic tissue/solid organ transplant
4. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
5. Evidence of interstitial lung disease.
6. cT4 tumor
7. Symptomatic acute cardiovascular or cerebrovascular disease
8. Known active HBV, HCV or HIV infection
9. Has any other active infection requiring systemic therapy.
10. Patients with active tuberculosis
11. Prior therapy with an anti-Programmed cell death protein 1 (anti-PD-1), anti-PD-L1, anti-Programmed cell death-ligand 2 (anti-PD-L2), anti-CD137 (4-1BB ligand, a member of the Tumor Necrosis Factor Receptor [TNFR] family), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
12. A diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
13. Patient has had a prior monoclonal antibody within 4 weeks prior to study Day 1
14. Patient has had prior chemotherapy, targeted small molecule therapy, or radiation therapy in history.
15. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
16. Has received a live vaccine within 30 days prior to the first dose of trial treatment. [Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines are live attenuated vaccines, and are not allowed.]
17. Has known hypersensitivity to pembrolizumab or any of the constituents of the product.
18. Other active malignancy requiring treatment Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
19. Lactating or pregnant women, women of child-bearing potential who do not agree to the usage of highly effective contraception methods (allowed methods of contraception, meaning methods with a rate of failure of less than 1% per year are implants, injectable contraceptives, combined oral contraceptives, intrauterine pessars (only hormonal devices), sexual abstinence or vasectomy of the partner). Women of childbearing potential must have a negative pregnancy test (serum β-hCG) at Screening.
20. Any psychiatric illness that would affect the patient's ability to understand the demands of the clinical trial
21. Patient has already been recruited in this trial
22. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.
23. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin E. Eichhorn, PD Dr. med., Principal Investigator — University Hospital Heidelberg
Locations (1):
- Universitätsklinikum Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi Y, Li J, Chen M, Liu H, Ma D, Lin Y, Wang M, Xu Y. Sarcoidosis-like reaction after neoadjuvant pembrolizumab combined with chemotherapy mimicking disease progression of NSCLC induced encouraging discovery of pathological complete response. Thorac Cancer. 2021 Dec;12(24):3433-3436. doi: 10.1111/1759-7714.14228. Epub 2021 Nov 11. PMID 34761878
- [Derived] Eichhorn F, Klotz LV, Kriegsmann M, Bischoff H, Schneider MA, Muley T, Kriegsmann K, Haberkorn U, Heussel CP, Savai R, Zoernig I, Jaeger D, Thomas M, Hoffmann H, Winter H, Eichhorn ME. Neoadjuvant anti-programmed death-1 immunotherapy by pembrolizumab in resectable non-small cell lung cancer: First clinical experience. Lung Cancer. 2021 Mar;153:150-157. doi: 10.1016/j.lungcan.2021.01.018. Epub 2021 Jan 21. PMID 33529989
- [Derived] Eichhorn F, Klotz LV, Bischoff H, Thomas M, Lasitschka F, Winter H, Hoffmann H, Eichhorn ME. Neoadjuvant anti-programmed Death-1 immunotherapy by Pembrolizumab in resectable nodal positive stage II/IIIa non-small-cell lung cancer (NSCLC): the NEOMUN trial. BMC Cancer. 2019 May 2;19(1):413. doi: 10.1186/s12885-019-5624-2. PMID 31046714

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 30
Completed | 29
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 60 [40 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 29
ECOG status [Count of Participants; unit: Participants] — Performance status according to the scoring system by the der Eastern Cooperative Oncology Group (ECOG), where patients scoring 0 and 1 are the most healthy:
  0 - Asymptomatic (Fully active, able to carry on all predisease activities without restriction)
  1 - Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work)
  Participants
    ECOG 0 | 14
    ECOG 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Treated in Compliance With Protocol
Description: The definition for this endpoint was neoadjuvant pembrolizumab treatment followed by successful curative intent tumor resection.
Time Frame: From screening until surgery, ca. 6-8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 29
Participants | 29

2. Primary Outcome: Tumor Response According to RECIST 1.1 Criteria
Description: Radiologic tumor assessments were performed at screening and pre-surgery.
Time Frame: From screening until pre-surgery radiologic assessment, ca. 6-8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 28
Participants
  Complete response | 0
  Partial response | 6
  Stable disease | 19
  Progressive disease | 3

3. Primary Outcome: Tumor Response Evaluation - Pathologic Response
Description: Pathologic regression grading according to Junker criteria.
  The following grades are defined:
  Grade I No tumor regression or only spontaneous tumor regression in the sections of the primary tumor and mediastinal lymph nodes.
  Grade IIa Morphological signs of therapy-induced tumor regression in the sections of the primary tumor and/or mediastinal lymph nodes: More than 10% vital tumor tissue
  Grade IIb Morphological signs of therapy-induced tumor regression: Less than 10% vital tumor tissue
  Grade III Complete tumor regression, no evidence of vital tumor in the sections of the primary tumor and/or mediastinal lymph nodes.
  Regression grades IIb and III suggest a good response to neoadjuvant therapy.
  Reference: Junker K, Langner K, Klinke F, Bosse U, Thomas M. Grading of tumor regression in non-small cell lung cancer : morphology and prognosis. Chest 2001; 120:1584-91.
Time Frame: From screening until surgery, ca. 6-8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 29
Participants
  Grade I | 4
  Grade IIa | 18
  Grade IIb | 3
  Grade III | 4

4. Primary Outcome: Tumor Response Evaluation - Δ Tumor Size
Description: Δ tumor size was defined as the difference [mm] between longest diameter at baseline and pre-surgery.
Time Frame: From screening until pre-surgery radiologic assessment, ca. 6-8 weeks
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 28
mm | -4.0 [-13.5 to 0.0]

5. Primary Outcome: Tumor Response - Δ PET Activity
Description: Δ PET activity (standardized uptake value [SUV]). This method uses radiolabeled tracer 82-deoxy-2-[18F]fluoro-D-glucose, FDG) during PET imaging of the tumor and accumulation of radiolabeled FDG measured by the PET scanner. Accumulation of FDG relative to normal tissue is related to the proliferative activity of malignant tissue and to the number of viable tumor cells. The endpoint is based on per-patient changes in tumor maximal standardized uptake value during PET examinations of the tumor before the start of treatment and after 2 cycles of neoadjuvant immunotherapy, i.e. between screening and shortly before surgery. Reduction of proliferative activity or of the number of viable tumor cells results in negative values.
Time Frame: From screening until pre-surgery radiologic assessment, ca. 6-8 weeks
Measure: Median (Inter-Quartile Range); unit: standardized uptake value [SUV]
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 28
standardized uptake value [SUV] | -1 [-7 to 2]

6. Secondary Outcome: Disease-free Survival at 6 Months
Description: Probability of disease-free survival (DFS) was calculated using Kaplan-Meier statistics from date of surgery to the date until tumor recurrence or death. Follow-up was until 24 months after last-patient-out.
Time Frame: 6 months after surgery, i.e. circa 8 months after treatment start
Measure: Number (95% Confidence Interval); unit: Probablity of DFS in %
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 29
Probablity of DFS in % | 86.2 [67.3 to 94.6]

7. Secondary Outcome: Disease-free Survival at 12 Months
Description: Probability of disease-free survival (DFS) was calculated from date of surgery until tumor recurrence or death using Kaplan-Meier statistics. Follow-up was until 24 months after last-patient-out.
Time Frame: 12 months after surgery, i.e. circa 14 months after treatment start
Measure: Number (95% Confidence Interval); unit: Probablity of DFS in %
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 29
Probablity of DFS in % | 86.2 [67.3 to 94.6]

8. Secondary Outcome: Overall Survival at 12 Months
Description: Probability of overall survival (OS) was calculated from date of surgery until date of death using Kaplan-Meier statistics. Follow-up was until 24 months after last-patient-out.
Time Frame: 12 months after surgery, i.e. circa 14 months after treatment start
Measure: Number (95% Confidence Interval); unit: Probability of OS in %
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 29
Probability of OS in % | 93.1 [75.1 to 98.2]

9. Secondary Outcome: Overall Survival at 18 Months
Description: as for outcome 8
Time Frame: 18 months after surgery, i.e. circa 20 months after treatment start
Measure: Number (95% Confidence Interval); unit: Probability of OS in %
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 29
Probability of OS in % | 89.7 [71.3 to 96.5]

10. Secondary Outcome: Overall Survival at 24 Months
Description: as for outcome 8
Time Frame: 24 months after surgery, i.e. circa 26 months after treatment start
Measure: Number (95% Confidence Interval); unit: Probability of OS in %
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 29
Probability of OS in % | 86.2 [67.3 to 94.6]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from signing of informed consent until 90 days after last dose of IMP (total: 20-22 weeks) or for 6 weeks after surgery (total: 12-14 weeks) if the subject initiated new anticancer therapy. Deaths were recorded for up to 26 months after treatment initiation.
Description: Note that deaths were recorded for up to 26 months after treatment initiation, but only for the purpose of collecting data for the overall survival efficacy endpoint. Of the total of 5 recorded deaths, only 1 fell within the time frame for safety reporting, and therefore, only 1 adverse event with fatal outcome is recorded in the safety database. This was a case of Acute Hepatic Failure reported as related to study treatment.
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 5/29
Serious Adverse Events (participants affected / at risk) | 8/29
Other Adverse Events (participants affected / at risk) | 21/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=29)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=29)
Autoimmune thyreoditis (Endocrine disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 4 (4)
Pain (General disorders) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3)
Decreased appetite (General disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3)
Paraesthesia (Nervous system disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT03197467/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT03197467/SAP_001.pdf